CLINICAL TRIAL: NCT03045627
Title: A Multi-center Randomized Open-label Clinical Trial of Ara-C, Aclarubicin Combined With PEG-G-CSF for Initial Treatment of Acute Myeloid Leukemia Patients
Brief Title: Clinical Trial of Ara-C, Aclarubicin Combined With PEG-G-CSF for Initial Treatment of AML Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AML- PEG-G-CSF
Record Dates: First submitted 2017-01-16; First posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; PEG-G-CSF
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Aclarubicin; pegylated granulocyte colony-stimulating factor, human; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Active Comparator): Ara-C, Aclarubicin Combined PEG-G-CSF
  ARA-C subcutaneously in a 12-hour infusion on days 1 through 14, Aclarubicin(Acla) 5～7mg/m2/d，intravenously on days 1 through 8, PEG-G-CSF 6mg subcutaneously on days 0. One course includes 28 days.
  Interventions: Drug: AraC; Drug: Aclarubicin; Drug: Peg-G-CSF
- Active comparator (Active Comparator): Ara-C, Aclarubicin Combined G-CSF
  ARA-C subcutaneously in a 12-hour infusion on days 1 through 14, Aclarubicin(Acla) 5～7mg/m2/d，intravenously on days 1 through 8, G-CSF 200 μg·m-2·d-1, subcutaneously on days 0 through 14. G-CSF was postponed or interrupted in case of white blood cell (WBC) count greater than 20 × 109/L .
  One course includes 28 days.
  Interventions: Drug: AraC; Drug: Aclarubicin; Drug: G-CSF

INTERVENTIONS:
Drug: AraC — ARA-C subcutaneously in a 12-hour infusion on days 1 through 14
  Other Names: cytarabine
Drug: Aclarubicin — Aclarubicin(Acla) 5～7mg/m2/d，intravenously on days 1 through 8
  Other Names: Aclarubicin A
Drug: Peg-G-CSF — PEG-G-CSF 6mg subcutaneously on days 0.
  Arms: Experimental
Drug: G-CSF — G-CSF 200 μg·m-2·d-1, subcutaneously on days 0 through 14.
  Arms: Active comparator

SUMMARY:
Most of patients with acute myeloid leukemia (AML) are elder and have poor prognosis despite induction chemotherapy.The regimen of cytarabine(Ara-C), aclarubicin and G-CSF (CAG regimen ) has been widely used in China for the treatment of acute myeloid leukemia (AML). Strategies to reduce the toxicity associated with intensive chemotherapy include the attenuated doses of standard regimens and myeloid growth factors. Granulocyte colony-stimulating factor(G-CSF) is efective in the prophylaxis and management of chemotherapy-induced neutropenia，but requires daily administration because of its short half-life． Pegylated granulocyte colony-stimulating factor (PEG-G-CSF )is a long-acting reagent that permits less frequent injection．The project is undertaken by Qilu Hospital of Shandong University and other well-known hospitals in China.In order to report the efficacy and safety of PEG-G-CSF combined with Ara-C and aclarubicin for the treatment of Acute Myeloid Leukemia, compared to the regimen of Ara-C, aclarubicin and G-CSF (CAG ).

DETAILED DESCRIPTION:
The Investigators are undertaking a parallel, multicentre, randomised open-label trial of newly diagnosed AML (not APL) patients in China. Participants are randomised selected to receive the regimen of Ara-C, aclarubicin and PEG-G-CSF , or the regimen of Ara-C, aclarubicin and G-CSF (CAG ).Platelet count, bleeding and other symptoms are evaluated before and after treatment. Adverse events are also recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. age 60 years and older, with an upper age limit of 75 years;
2. diagnosis of AML other than APL
3. Adequate hepatic and renal function (aspartate aminotransferase [AST], alanine aminotransferase [ALT], bilirubin and creatinine < 2.5 x upper normal limit).

Exclusion Criteria:

1. History of severe congestive heart failure or other cardiac disease that contraindicates the use of anthracyclines, including idarubicin
2. Use of recreational drugs or history of drug addiction, within the prior 6 months
3. Known history of positive hepatitis B surface antigens or hepatitis C virus (HCV) antibodies
4. Patients with documented cases of human immunodeficiency virus (HIV)

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Complete remission (CR) | 60 days from the enrollment
  Bone marrow blasts not more than 5%, absence of blasts with Auer rods, absence of extramedullary disease, absolute neutrophil count more than 1*10^9/L, platelet count more than 100*10^9/L,independence of red cell transfusions

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hospital, Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided